CLINICAL TRIAL: NCT06368102
Title: Prophylactic Effects of Different Duration of Intravenous Ampicillin for Preventing Surgical Site Infection in Third Molar Surgery: a Randomized Controlled Trial
Brief Title: Prophylactic Effects for Preventing Surgical Site Infection in Third Molar Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Uji Takeda Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R6-03
Record Dates: First submitted 2024-04-10; First posted 2024-04-16 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Ampicillin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 1day-group (Experimental): Participants will receive 1g of IV ampicillin before surgery and 1 time after surgery on the day of surgery (total 2g)
  Interventions: Drug: Ampicillin
- 2day-group (Experimental): Participants will receive 1g of IV ampicillin before surgery and 2 times after surgery up to the next day (total 3g)
  Interventions: Drug: Ampicillin

INTERVENTIONS:
Drug: Ampicillin — Total 2g vs 3g

SUMMARY:
The purpose of this study is to determine the incidence of surgical site infection (SSIs) after third molar surgery for different duration of intravenous ampicillin administration.

DETAILED DESCRIPTION:
In recent years, the increase in drug-resistant bacteria and associated infections has become one of the major issues in the international community as adverse events associated with the inappropriate use of antimicrobial agents. Although the frequency and percentage of inappropriate use is currently unknown, it has been shown that at least 30% of antimicrobials prescribed in the U.S. are inappropriately used. If no action is taken against inappropriate antimicrobial use, it is estimated that 10 million people will die annually worldwide from drug-resistant organisms by 2050, with an estimated 4.9 million deaths related to drug-resistant organisms and 1.2 million deaths due to drug-resistant organisms already estimated for 2019. In addition, while the development of new antimicrobial agents has declined since the 1980s, the threat of new drug-resistant organisms, especially in hospitals, has increased, and if antimicrobial agents are not used appropriately, there is concern that there will be no effective antimicrobial agents available to treat infections in the future. It is important to avoid such situations by using antimicrobial agents, which are a limited resource, appropriately at this stage, and appropriate use of antimicrobial agents is necessary to prevent drug resistance (Antimicrobial Resistance: AMR).

Third molar extraction is the most commonly performed procedure in oral and maxillofacial surgery. One of the main complications after third molar extractions is surgical site infection (SSIs), which is reported to manifest as swelling, pain, abscess, and fever. According to a Cochrane review of randomized controlled trials, the risk of SSIs after third molar extraction in physically fit young patients is about 10%, but in patients with low immunity before extraction, the risk increases up to 25%. Prophylactic administration of antimicrobial agents has an important role in preventing SSIs. However, the efficacy of antimicrobial prophylaxis against SSIs in third molar extractions is controversial. While some studies have reported that antimicrobials are effective in preventing SSIs after third molar extraction, others have reported that they are not.

Guidelines for third molar extraction vary widely in the duration of antimicrobial administration (e.g., Japanese guidelines state a single dose to within 48 hours). In clinical practice, the final decision lies with the surgeon, but this difference in dosing period is a source of confusion. If the duration of administration could be shortened without increasing SSIs, it would contribute to the current presentation of AMR. Therefore, the purpose of this study is to examine the effect of different durations and doses of penicillins, which are considered first-line drugs after third molar surgery, on the prevention of SSIs.

ELIGIBILITY:
Inclusion Criteria:

* Minimum age of 20 years
* American Society of Anesthesiologists (ASA) physical status of 1
* Planned extraction of bilateral mandibular third molar with the necessity of bone removal based on panoramic radiography in an inpatient setting under IV sedation
* Agreement to follow the study protocol

Exclusion Criteria:

* Pregnancy or suspicion of pregnancy
* Allergy and/or contraindication to ampicillin
* History of a known SSI risk factors, such as diabetes, steroid or immunosuppressant use, and endocarditis
* Receiving any antibiotic therapy
* Active infection of the third molars with pus, edema, and trismus

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2025-08-01 (Actual); Study Completion 2025-09-01 (Actual)

PRIMARY OUTCOMES:
Occurrence of surgical site infection | 30 days
  is evaluated based on the guidelines by the Center for Disease Control and Prevention (CDC) and Clavien-Dindo classification system: within 30 days postoperatively, drainage from a surgical wound or abscess, requiring treatment with antimicrobial agents.

SECONDARY OUTCOMES:
Occurrence of alveolar osteitis | 7 days
  is evaluated based on the postoperative pain within and around the extraction site with increasing severity accompanied by partially or completely collapsed clots in the alveolar fossa, and the presence of halitosis

CONTACTS AND LOCATIONS:
Overall Officials: Keita Kano, PhD, Study Chair — Uji Takeda Hospital
Locations (1):
- Uji Takeda Hospital, Uji, Japan